CLINICAL TRIAL: NCT04258332
Title: Dietary Sodium Inflammation and Salt Sensitivity of Blood Pressure
Brief Title: CARDIA-Salt Sensitivity of Blood Pressure (SSBP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Northwestern University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Deepak Gupta, Asst Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 190622
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Salt Sensitivity of Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Salt Diet then Low Salt Diet (Other): The high-salt diet will be achieved through the supplementation of each participant's usual diet with Na+ bullion packets (2 packets per day). This will increase Na+ intake by approximately 2,200 mg (≈100 mEq Na+) to a total greater than 5,000 mg Na+ per day based on prior estimates of Na+ intake (see section C1.2). In addition, 1,000 mg of calcium carbonate (provided via Tums tablets) will be taken daily on the high Na+ diet to reduce the potential impact of changes in calcium intake on blood pressure.
  The low-salt diet is comprised of 7 days of freshly prepared frozen meals, snacks, and Na+ free water. All low-salt meals will be prepared in each site's Metabolic Kitchen, with standardization of diets across sites. The low-salt diet includes: 20 mEq Na+ (±2 mEq) (460 mg/day), 100 mEq potassium (±2 mEq), and 1,000 mg calcium (±50 mg).
  Interventions: Dietary Supplement: High Salt Diet; Dietary Supplement: Low Salt Diet
- Low Salt Diet then High Salt Diet (Other): The low-salt diet is comprised of 7 days of freshly prepared frozen meals, snacks, and Na+ free water. All low-salt meals will be prepared in each site's Metabolic Kitchen, with standardization of diets across sites. The low-salt diet includes: 20 mEq Na+ (±2 mEq) (460 mg/day), 100 mEq potassium (±2 mEq), and 1,000 mg calcium (±50 mg).
  The high-salt diet will be achieved through the supplementation of each participant's usual diet with Na+ bullion packets (2 packets per day). This will increase Na+ intake by approximately 2,200 mg (≈100 mEq Na+) to a total greater than 5,000 mg Na+ per day based on prior estimates of Na+ intake (see section C1.2). In addition, 1,000 mg of calcium carbonate (provided via Tums tablets) will be taken daily on the high Na+ diet to reduce the potential impact of changes in calcium intake on blood pressure.
  Interventions: Dietary Supplement: High Salt Diet; Dietary Supplement: Low Salt Diet

INTERVENTIONS:
Dietary Supplement: High Salt Diet — Patients will be randomized to be on a high salt diet for 7 days.
Dietary Supplement: Low Salt Diet — Patients will be randomized to be on a low salt for 7 days.

SUMMARY:
Salt sensitivity of blood pressure (SSBP) is defined as the change in blood pressure (BP) in relation to change in salt intake. An increase in BP from low- to high-salt diet is common and associated with an increased risk of cardiovascular morbidity and mortality, even among normotensive individuals. Yet, the pathophysiology of SSBP is not well understood. The prevailing paradigm is that abnormalities of neurohormones that regulate sodium (Na+) retention and excretion and/or Na+ transporting pathways create Na+ imbalances that underlie susceptibility to SSBP. As a homeostatic mechanism, BP fluctuates to maintain Na+ balance, i.e. higher BP is needed for pressure natriuresis to excrete excess Na+. An alternate framework emphasizes vascular dysregulation as the inciting mechanism. In both constructs, how Na+ itself influences BP remains incompletely understood. Our preliminary work suggests that excess Na+ induces a pro-inflammatory state that sustains higher BP. Interleukin-6 (IL-6) drives the induction of interleukin-17 (IL-17) secreting T helper 17 cells that were recently demonstrated to be pathogenic in response to Na+ exposure. IL-6, IL-17 and related cytokines regulate renal Na+ transporters and raise BP through vascular inflammation, fibrosis, and impaired vasodilation. The immune response to high- and low-salt diet in humans, however, is not completely understood, emphasizing the need for more detailed human studies, with deeper immune profiling under controlled salt conditions and with neurohormonal assessment. Our overarching postulate is that the inflammatory response to excess dietary salt intake is associated with SSBP. The Coronary Artery Risk Development in Young Adults (CARDIA) study is the ideal cohort in which to translate our preliminary findings. Investigators propose to investigate SSBP in CARDIA using standardized low- and high-salt diets and 24-hour ambulatory BP monitoring. Investigators will quantify SSBP in a total of 500 participants from the Chicago and Birmingham field centers during the upcoming year 35 exam (beginning in 2020). Our specific aims are: 1) to define the distribution of SSBP and its clinical correlates in a contemporary community-based US cohort of middle-aged individuals; 2) to investigate the immune response to dietary salt loading, and 3) to investigate the association between the immune and BP responses to dietary salt loading. The proposed study represents a unique opportunity to leverage a large, well-phenotyped cohort to test novel hypotheses regarding SSBP. Phenotyping SSBP using standardized high- and low-salt diets in CARDIA will be novel as this has never been performed in any of the existing US based NHLBI sponsored cardiovascular epidemiologic cohorts. The proposed work has the potential to yield a more readily available approach for differentiating an individual as salt-sensitive or resistant. New insights into the pathophysiology of SSBP should also provide a foundation for investigating high-impact clinical applications, by informing future studies of therapies directed at SSBP. The scientific rigor is further enhanced by the rich clinical, genetic, and biochemical data available in CARDIA.

ELIGIBILITY:
Inclusion Criteria:

Potentially eligible individuals must consent to and be willing to adhere to the study protocol. We will include individuals not taking anti-HTN medications, i.e. normotensives and untreated hypertensives, and individuals with controlled HTN by use of ≤ 3 anti-HTN medications.

Exclusion Criteria:

* Unwilling to adhere to the study protocol
* Resistant HTN, defined as taking ≥ 4 anti-HTN medications to control BP or uncontrolled BP despite ≥ 3 anti-HTN medications that includes a diuretic
* Contraindications to high- or low-salt diet (e.g. heart, renal, or liver failure, postural orthostatic tachycardia syndrome)
* Use of salt tabs, fludricortisone, midodrine
* Contraindications to 24hr ABPM: bilateral upper extremity lymphedema, cuff will not fit
* Medical contraindications to foods, e.g. celiac disease, nut allergy, egg allergy, etc.
* Year 35 core exam systolic BP < 90 or > 160 mm Hg or diastolic BP < 50 or > 100 mm Hg
* Current use of steroids, NSAIDS, anti-inflammatories
* Rheumatologic condition (e.g. Lupus, Rheumatoid Arthritis, Psoriatic arthritis, Inflammatory Bowel Disease, Multiple Sclerosis
* Immune deficiency or immunosuppressed

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Salt sensitivity of blood pressure | 14 days
  The change in 24-hour ambulatory mean arterial pressure (MAP) from one week of high-salt to one week of low-salt diet
Immune response to dietary salt loading, IL-6 | 14 days
  Circulating levels of IL-6
Immune response to dietary salt loading, Change in circulating levels of IL-17 | 14 days
  Circulating levels of IL-17
Immune response to dietary salt loading, IL-10 | 14 days
  Circulating levels of IL-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Research data will be shared according to the most recent NIH guideline. The data collected will be made available by the CARDIA Data Coordinating Center (DCC) both to the study for use by other investigators and to NHLBI for inclusion in the NHLBI's Data Repository Program, in accordance with the NHLBI Policy for Data Sharing from Clinical Trials and Epidemiological Studies, http://www.nhlbi.nih.gov/funding/datasharing.htm. Through the conduct of the study and in resource sharing, attention will be given to protect private health information; thus, we will make data available to others through the CARDIA DCC under a data use agreement specifying (1) to use the data only for research purposes and not to identify an individual participant; (2) to secure the data using appropriate computer technology; and (3) to destroy or return the data after analyses are completed. The overall CARDIA DCC at the UAB will be responsible for overseeing approval and sharing of research data.

REFERENCES:
- [Derived] Gupta DK, Lewis CE, Varady KA, Su YR, Madhur MS, Lackland DT, Reis JP, Wang TJ, Lloyd-Jones DM, Allen NB. Effect of Dietary Sodium on Blood Pressure: A Crossover Trial. JAMA. 2023 Dec 19;330(23):2258-2266. doi: 10.1001/jama.2023.23651. PMID 37950918

DOCUMENTS (1):
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT04258332/ICF_000.pdf